CLINICAL TRIAL: NCT06660498
Title: Pomalidomide as an Immune-enhancing Agent for the Control of HIV (PEACH): An Investigator-initiated Phase I/IIb Clinical Trial in People Living With HIV on ART and During Analytical Treatment Interruption
Brief Title: Pomalidomide as an Immune-enhancing Agent for the Control of HIV
Acronym: PEACH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-512797-10-00 (EU CT no.)
Record Dates: First submitted 2024-10-07; First posted 2024-10-28 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-09

CONDITIONS: HIV-1 Infection
Keywords: Immune-enhancing therapy; HIV; ART; Analytical treatment interruption; Investigator-initiated
MeSH Terms: interventions — pomalidomide; Aspirin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to pomalidomide 2 mg/d or matching placebo concurrent with aspirin 75 mg.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pomalidomide (Active Comparator): This arm will receive pomalidomide 2 mg oral capsules
  Interventions: Drug: Pomalidomide 2 mg; Drug: Aspirin 75 mg
- Placebo (Placebo Comparator): This arm will receive placebo (oral capsules with no active drug)
  Interventions: Drug: Placebo; Drug: Aspirin 75 mg

INTERVENTIONS:
Drug: Pomalidomide 2 mg — Participants will receive pomalidomide 2 mg/d concurrently with aspirin 75 mg for three cycles, each consisting of 21 days on and a minimum of 7 days off.
  Arms: Pomalidomide
Drug: Placebo — Participants will receive placebo concurrently with aspirin 75 mg for three cycles, each consisting of 21 days on and a minimum of 7 days off.
  Arms: Placebo
Drug: Aspirin 75 mg — Auxiliary Medicinal Product

SUMMARY:
This study is designed to evaluate the safety and efficacy of pomalidomide in HIV-1-infected individuals on ART and to determine the impact of pomalidomide on virological control in people living with HIV during an analytical treatment interruption.

ELIGIBILITY:
Documented HIV-1 infection

* Age 18-70 years, both included.
* Receiving combination ART for at least 1 year and being on the same ART regimen for at least 4 weeks at the screening visit
* HIV-1 plasma RNA <50 copies/mL for >1 year and <20 copies/mL at screening. Episodes of a single HIV plasma RNA >50-500 copies/mL will not exclude participation if the subsequent HIV plasma RNA was <50 copies/mL
* CD4+ T cell count >500 cells/uL at screening
* Ability and willingness to provide informed consent and to continue ART throughout the study phase I and to discontinue ART at the commencement of study phase II.
* All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) during the study.
* A female participant, may be eligible to enter and participate in the study if she:

  * Is of non-child-bearing potential defined as either:

    * Age ≥ 50 years and naturally amenorrheic for ≥ 1 year (amenorrhoea following cancer therapy or during breast-feeding does not rule out childbearing potential)
    * Premature ovarian failure confirmed by a specialist gynecologist
    * Previous bilateral salpingo-oophorectomy, or hysterectomy
    * XY genotype, Turner syndrome, uterine agenesis
  * Is of child-bearing potential with a negative pregnancy test at both Screening and Day 0 and agrees to use one of the following methods of contraception to avoid pregnancy:

    * Complete abstinence from penile-vaginal intercourse from 4 weeks prior to administration of investigational medical product (IMP), throughout the study, and for at least 4 weeks after discontinuation of all study medications
    * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year
    * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject
    * Approved hormonal contraception (Where other medications to be used in the study (e.g., efavirenz and darunavir) are known, or are likely, to significantly interact with systemic contraceptives, resulting in decreased efficacy of the contraceptive, then alternative methods of non-hormonal contraception are recommended)
    * Any other method with published data showing that the expected failure rate is <1% per year
    * Any contraception method must be used consistently, in accordance with the approved product label and for at least 4 weeks after discontinuation of study therapy.

A heterosexually active male participant, may be eligible to enter and participate in the study if he is:

* Willing to complete abstinence from penile-vaginal intercourse from 4 weeks prior to administration of IP, throughout the study, and for at least 4 weeks after discontinuation of all study medications
* willing to use an effective method of contraception (condom) including those who have had vasectomy performed
* agree on the use of an effective method of contraception with an effective failure rate of <1% by his partner (hormonal contraception, intra-uterine device (IUD), or anatomical sterility) from the day prior to the first dose and for at least 4 weeks after discontinuation of study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment, measured as the time from ART cessation until meeting ART restart criteria. | From ATI to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
Safety of treatment, measured by the number of treatment-emergent adverse events (AEs) of grade 3 or higher that are probably or definitely related to the study treatment. | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria

SECONDARY OUTCOMES:
Safety, defined as all other treatment-emerging adverse events (AEs) | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
  AEs are graded according to severity and assessed as either not related or possibly, probably or definitely related to study treatment.
Rebound viral kinetics during the ATI, including plasma HIV-1 RNA copies/mL doubling times | From ATI to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
The proportion of participants maintaining HIV-1 RNA levels below 1,000 copies/mL at the end of the ATI. | From ATI to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
The proportion of participants who have not met ART restart criteria at the end of the ATI. | From ATI to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
The frequency of peripheral blood CD4+ T cells containing total and intact HIV-DNA while on suppressive ART | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
HIV-specific CD4+ responses | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
HIV-specific CD8+ T cell responses | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
The proportion of cells containing constitutive and inducible MS HIV-RNA | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
The level of CA-US HIV RNA in peripheral blood CD4+ T cells | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
Numbers of B cells, total lymphocytes, CD8+ T cells and CD4+ T cells including memory subsets | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria
Proportions of B cells, total lymphocytes, CD8+ T cells and CD4+ T cells including memory subsets | From enrollment to the end of treatment at visit 18 or 16 weeks after meeting ART restart criteria

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Rasmussen, Associate professor, MD, PhD, Principal Investigator — University of Aarhus
Locations (2):
- Royal Melbourne Hospital, Melbourne, Australia
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The participant data will be shared with collaborative researchers but in an anonymous form that cannot be traced to the individual participant, according to the General Data Protection Regulation (GDPR) of the European Union.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2024-September 2026
Access Criteria: Since the study was approved in September 2024, there has been open access to the study protocol, the statistical analysis plan, and the informed consent form through the CTIS platform.